CLINICAL TRIAL: NCT04958356
Title: Newborn Screening for Genetic Susceptibility to Type 1 Diabetes and Celiac Disease and Prospective Follow-up Study
Acronym: BABYSCREEN
Status: Active, not recruiting | Type: Observational
Sponsor: University of Helsinki (Other)
Responsible Party: Principal Investigator, Mikael Knip, Professor, Research Director, University of Helsinki
Other Study IDs: 728/2018
Record Dates: First submitted 2019-02-27; First posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Type1diabetes; Celiac Disease
Keywords: type 1 diabetes; celiac disease
MeSH Terms: conditions — Celiac Disease; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples Without DNA — EDTA sample from cord blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with increased risk for T1D and/or CeD: The participants carrying HLA-conferred susceptibility to type 1 diabetes will be screened annually for four diabetes predictive autoantibodies and followed up to 1-3 years of age. The participants carrying HLA-conferred susceptibility to celiac disease are screened for tissue transglutaminase antibodies (tTGA) at the age of 1 and 3 years. If a child tests positive for such autoantibodies, endomysial antibodies will be analyzed.

SUMMARY:
This is an observational study, in which newborn infants from the general population are screened at birth for HLA-conferred susceptibility to type 1 diabetes and celiac disease. The participants carrying genetic susceptibility to type 1 diabetes (approximately 9.5%) will be analyzed for diabetes-associated autoantibodies at the age of 1, 2 and 3 years, while those predisposed to celiac disease (about 14%) will be screened for tissue transglutaminase antibodies at the age of 1 and 3 years. The intention is to screen annually 10,400 newborn infants for a period of 3 years. About 988 infants are each year identified as a child at risk for type 1 diabetes, and it is expected that around 80% of the families with such a child are willing to join the autoantibody screening. Approximately 1456 infants are each year recognized as a child at risk for celiac disease, and again the expectation is that 80% of the families will join the antibody screening program.

DETAILED DESCRIPTION:
The aim of the BABYSCREEN project is to identify newborn infants with HLA-conferred susceptibility to T1D and/or CeD from the general population and to observe such children for the appearance of disease-associated autoantibodies and clinical disease up to the age of 1-3 years. The plan is to screen all infants with maternal consent born in one of the two delivery hospitals in the metropolitan Helsinki area, i.e. Women's Hospital in Helsinki and Jorvi Hospital in Espoo. The parents to be will be informed about the study and invited during pregnancy to take part in the study after the birth of their baby. The pregnant woman is asked to give her electronic consent to participation through the Women's website (https://www.terveyskyla.fi/naistalo) or a written informed consent on paper after both parents have acquainted themselves with the study. The only inclusion criterion will be informed consent signed by the mother.

The screening activity will be carried out over a 3-year period. The annual number of births in the Helsinki region is about 13,000. It is expected that at least 80% of the parents will give their informed consent to participation in the study. Accordingly about 31,200 newborn infants would be screened for genetic susceptibility to T1D and CeD. The following HLA genotypes represent those predisposing to T1D: (i) the high-risk genotype (DR3)-DQA1*05-DQB1*02/DRB1*04:01/2/4/5;)-DQA1*03-DQB1*03:02; (ii) the moderately increased-risk genotype DRB1*04:01/2/5-DQA1*03-DQB1*03:02/neutral haplotype; (iii) the slightly increased-risk genotype (DR3)-DQA1*05-DQB1*02/ (DR9)-DQA1*03-DQB1*03:03; (iv) DR4 homozygosity DRB1*04:01/2/4/5)-DQA1*03-DQB1*03:02/DRB1*04:01/2/4/5)-DQA1*03-DQB1*03: 02; and (v) DR3 homozygosity (DR3)-DQA1*05-DQB1*02/(DR3)-DQA1*05-DQB1*02. To cover those with genetic susceptibility to CeD also all other genotypes including the DR3-DQ2 haplotype will be identified. Their proportion among Finnish infants is 14%. This screening protocol identifying 23.5% of the screened infants as at-risk children has a sensitivity of 64.6% for T1D and more than 90% for CeD. Around 9.5% will carry HLA susceptibility to T1D and an additional 14% predisposition to CeD. With an expected consent rate of 80%, approximately 988 participants with HLA-defined predisposition to T1D (about 370 of them having also susceptibility to CeD) and 1,456 participants with HLA-conferred susceptibility to only CeD would be ended up each year. In addition, DNA will later be extracted from cord blood to identify genes outside the HLA gene region conferring increased risk for T1D and/or CeD.

Families with a baby carrying a predisposing HLA genotype are invited to follow-up for the appearance of predictive autoantibodies. The participants genetically at risk for T1D will be screened with the guardians' consents annually for four diabetes predictive autoantibodies and followed up to 1-3 years of age. If a participant tests positive for one or more autoantibodies at a given age, he/she will be invited for a second sample within 2 months from the first positive sample. If a child test positive for multiple (≥ 2) autoantibodies, HbA1c will be analyzed and an oral glucose tolerance test carried out to diagnose or exclude dysglycemia. Dysglycemic participants will be referred to a pediatric unit taking care of children with T1D for continued monitoring.

The participants at risk for CeD are screened for tissue transglutaminase antibodies (tTGA) at the age of 1 and 3 years. If a child tests positive for such autoantibodies, endomysial antibodies will be analyzed. Children testing positive for both autoantibodies will be referred to a pediatríc gastroenterologist for consultation.

One objective of this project is to prevent diabetic ketoacidosis in those participants who progress to clinical T1D and to diagnose early the development of CeD to prevent its complications. This serves also as a demonstration project for the potential benefits achieved with early population-based screening of two common chronic childhood disorders.

The following information will be collected from the participants in the screening study; gestational age, route of delivery, gender, birth weight and length, head circumference, and Apgar score. In addition, information on autoimmune diseases in family will be collected at the beginning of the study and at the last study visit by electronic questionnaire, since any autoimmune disease in the family increases the risk of T1D and/or CeD in other family members. Growth will be monitored in the participants in the follow-up study.

Those at risk for T1D will be screened annually for the four biochemical autoantibodies predicting T1D, i.e. insulin autoantibodies (IAA) and antibodies to glutamate decarboxylase GADA), islet antigen 2 (IA-2A) and zinc transporter 8 (ZnT8A). These autoantibodies are analyzed with specific radiobinding assays. If a participant tests positive for one or more autoantibodies at a given age, he/she will be invited for a second sample within 2 months from the first positive sample. Participants with confirmed positivity for multiple (≥2) autoantibodies, will be invited for a new visit for assessing possible signs of dysglycemia. A HbA1c sample is taken and a 2-hour oral glucose tolerance test will be carried out. If the child has signs of dysglycemia, he/she will be referred to a pediatric unit taking care of patients with T1D for contínued follow-up. Participants with confirmed positivity for T1D associated autoantibodies at the last follow-up sample, will be invited to come to a new visit for assessing T1D associated autoantibodies after 3 years.

The children predisposed to CeD will be analyzed for IgA and IgG class tTGA at the age of 1 or 1 and 3 years of age. If the child tests unequivocally positive for tTGA, the positive sample will be analyzed for endomysial antibodies. If the participant has both autoantibodies, she/he will be referred to a pediatric gastroenterologists for consideration of duodenal biopsy. Participants with confirmed positivity for tTGA at the last follow-up sample, will be invited to come to a new visit for assessing CeD associated autoantibodies after 3 years.

ELIGIBILITY:
Inclusion Criteria:

* mother has given an informed consent

Exclusion Criteria:

-

Ages: 1 Minute to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Delivery hospitals in the Helsinki region. The number of annual births is approximately 13,000. Close to half of the newborn infants will be girls. The investigators expect that around 80% of the families (10,400) will give their informed consent to the genetic screening of their infant. About 9.5% of the infants screened (n=988) will carry HLA-conferred susceptibility to type 1 diabetes and approximately 14% (n=1456) predisposition to celiac disease. The families with at-risk infants will be invited to the autoantibody follow-up to the age of 3 years.
Sampling Method: Probability Sample
Enrollment: 9690 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with confirmed positivity for at least one diabetes-associated autoantibody (insulin autoantibodies and antibodies to GAD65, islet antigen 2 and zinc transporter 8) or confirmed positivity for tissue transglutaminase antibodies | December 31, 2022
  Antibodies listed in the title are analyzed by specific radiobinding assays. The cut-off limit of antibody positivity is defined based on 350 healthy children. Confirmed positivity refers to positive test results in at least two sequential samples. The autoantibodies are analyzed at the age of 1, 2 and 3 years. If a child tests positive, the result will be confirmed in a second sample taken within 2 months after the initially positive sample. The autoantibody screening allows the identification of participants who will present with preclinical or clinical disease before the age of 3 years. This will minimize the frequency of diabetic ketoacidosis among those participants, who progress to clinical T1D. Untreated CeD is associated with health sequelae. Early diagnosis of celiac disease based on screening for genetic disease susceptibility at birth combined with follow-up for the appearance of disease predictive autoantibodies will effectively prevent such problems.

CONTACTS AND LOCATIONS:
Overall Officials: Mikael Knip, MD, Principal Investigator — University of Helsinki
Locations (1):
- Hospital District of Helsinki and Uusimaa, Helsinki, HUS, Finland

IPD SHARING:
Plan to Share IPD: No